CLINICAL TRIAL: NCT06650891
Title: The Adjunctive Effect of Quercetin on Postoperative Pain Management Following Cesarean Section
Brief Title: Quercetin Effect on Post-ceserean Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Nouran Omar El Said, Lecturer in. Pharmacy Practice & Clinical Pharmacy, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RFC-PH-3/2024
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Post Operative Pain; Cesarean Section Complications
Keywords: post-operative pain; Cesarean section; quercetin; opioid use
MeSH Terms: conditions — Pain, Postoperative | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quercetin (Experimental): receive 500mg of oral quercetin 1 hour preoperatively.
  Interventions: Drug: Quercetin
- Placebo (Placebo Comparator): receive placebo 1 hour preoperatively
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Quercetin — oral quercetin prior to surgery
  Arms: Quercetin
Other: Placebo — capsule identical looking to quercetin
  Arms: Placebo

SUMMARY:
The cesarean section is a common gynecological surgery, requiring effective pain management to prevent complications and immobility. Inadequate pain control can lead to longer hospital stays, higher readmission rates, and dissatisfaction with healthcare. Traditional analgesics, such as opioids, have proven effective in alleviating pain, but they can cause side effects. Therefore, researchers are exploring compounds that can reduce opioid analgesic needs and improve pain control. Quercetin has anti-nociceptive effects in rodent models of chronic pain, including inflammatory, neuropathic, and cancer pain. There are limited clinical studies on the effect of quercetin on acute or chronic pain. The current study is designed to assess the efficacy of preoperative quercetin administration in acute post-operative pain following cesarean section.

DETAILED DESCRIPTION:
The cesarean section is a common gynecological surgery, accounting for 40-50% of deliveries in public hospitals. Effective pain management following a cesarean delivery is crucial, as inadequate control can hinder a mother's capacity to care for her newborn. Uncontrolled postoperative pain can lead to patient immobility, increasing the risk of thromboembolic complications. Failure to adequately manage pain can result in economic and medical issues, including longer hospital stays, higher readmission rates, increased patient recovery costs, and patient dissatisfaction with the quality of healthcare provided.

Opioid medications, particularly when administered via injection, have proven effective in alleviating acute pain, but they are associated with dose-related side effects. Therefore, it is prudent to investigate compounds that can potentiate the analgesic effects of opioids, enabling improved pain control while minimizing opioid consumption. Quercetin, a flavonoid and polyphenol found in various plants and fruits, has been studied for its anti-inflammatory, free radical scavenging, antidiabetic, anticancer, cardiovascular, hepatoprotective, neuroprotective, antiplatelet, antibacterial, and anti-obesity effects. Recent evidence indicates quercetin possesses anti-nociceptive effects in rodent models of chronic pain, including inflammatory pain, neuropathic pain, and cancer pain.

Quercetin has great potential for clinical use in pain treatment, as its safety is well established. However, there are limited clinical studies on the effect of quercetin on acute or chronic pain. The current study aims to assess the efficacy of preoperative quercetin administration in acute post-operative pain following cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Referred to elective (non-emergency) cesarean section
* Undergoing spinal anesthesia) with American Society of Anesthesiologists (ASA) classification I and II
* Term gestational age

Exclusion Criteria:

* History of seizures
* Pre-eclampsia or eclampsia
* Hypertension
* Use of narcotic painkillers for 24 h before the intervention
* Medications inducing neuropathy including Amiodarone, Metronidazole, Phenytoin & Colchicine.
* Prolongation of cesarean section (more than 1.5 h)
* Increase in the size of the incision
* Occurrence of any unusual complication during surgery,
* Failure of spinal anesthesia and its conversion to general anesthesia
* Contraindications to spinal anesthesia
* Use of interacting medication: fluoroquinolones, loratadine, fexofenadine, alvimopan, armodafinil

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Pain intensity (2 hours) | 2 hours
  Pain intensity using 10 cm Visual analog scale (VAS) scale
Pain intensity (6 hours) | 6 hours
  Pain intensity using 10 cm Visual analog scale (VAS) scale
Pain intensity (12 hours) | 12 hours
  Pain intensity using 10 cm Visual analog scale (VAS) scale
Pain intensity (24 hours) | 24 hours
  Pain intensity using 10 cm Visual analog scale (VAS) scale

SECONDARY OUTCOMES:
Nausea & vomiting (2 hours) | 2 hours
  severity of nausea/vomiting (n/v) using a numerical scale from 0 to 2 (0 = no nausea, 1 = mild n/v, and 2 = severe n/v)
Nausea & vomiting (6 hours) | 6 hours
  severity of nausea/vomiting (n/v) using a numerical scale from 0 to 2 (0 = no nausea, 1 = mild n/v, and 2 = severe n/v)
Nausea & vomiting (12 hours) | 12 hours
  severity of nausea/vomiting (n/v) using a numerical scale from 0 to 2 (0 = no nausea, 1 = mild n/v, and 2 = severe n/v)
Nausea & vomiting (24 hours) | 24 hours
  severity of nausea/vomiting (n/v) using a numerical scale from 0 to 2 (0 = no nausea, 1 = mild n/v, and 2 = severe n/v)
Rescue analgesia | 24 hours
  The patient's first request for postoperative analgesia
Opioid intake | 24 hours
  The patient's opioid intake in the 24-h after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- El Matarya Teaching Hospital,, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed Elmokadem E, Khaled Abou El Fadl D, Bassiouny AM, Mahmoud MMAE, Samy M, El Said NO. The Adjunctive Effect of Quercetin on Postoperative Pain Management Following Cesarean Section: A Randomized Controlled Study. Drug Des Devel Ther. 2025 Jul 14;19:6009-6024. doi: 10.2147/DDDT.S526188. eCollection 2025. PMID 40687903